CLINICAL TRIAL: NCT02209142
Title: Blood Biomarkers in Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-19
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Major Depressive Disorder
Keywords: Major depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pan-genomic screen (Experimental): A pan-genomic screen by blood prelevement and psychometric data collection will be set-up on a subset of MDE and control samples to identify mRNA candidates for a transcriptional signature of MDE,
  Interventions: Other: blood prelevement; Other: psychometric data collection
- control (Sham Comparator): a pan genomic screening by blood prelevement and psychometric data collection wil be performed on healthy subject
  Interventions: Other: blood prelevement; Other: psychometric data collection

INTERVENTIONS:
Other: blood prelevement — blood sample will be done at the inclusion then at T 2 weeks, T8 weeks, T30weeks
Other: psychometric data collection
  Other Names: psychometric data collection wil be done ( hamilton scale and clinical exam)

SUMMARY:
Depression is a leading cause of disability worldwide, affecting nearly 16% of the general population. Its physiopathology remains unclear. Based on gene-environment studies and epigenetic studies, a main hypothesis proposed that the major depressive episode (MDE) results from the convergence of multiple factors including biological factors such as multi-genic vulnerability, hormonal and immunological variations as well as environmental factors. As a consequence, mRNA could define a biological signature of the MDE.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder at inclusion according to the DSM IV at the time of the inclusion,

  * Having a score on the scale of depression of Hamilton ( HDRS-17) > 19 at the time of the inclusion,
  * Taken care by a grown-up psychiatric department, that the coverage(care) is realized in ambulatory or during a hospitalization

Exclusion Criteria:

* Schizophrenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
describe a transcriptional signature of the Major Depressive Episode. | 6 months
  The major aim of our study is to compare the expression level of selected genes between patient suffering from major depression and control subjects and within patients across the MDE evolution. We plan to describe a transcriptional signature of the MDE.

SECONDARY OUTCOMES:
evaluate the role played by confounding factors as genetic polymorphisms, | 6 months
  evaluate the role played by confounding factors as genetic polymorphisms to distinguish bipolar from unipolar depression

OTHER OUTCOMES:
evaluate the role played by confounding factors as immune phenotype | 6 months
  evaluate the role played by confounding factors as immune phenotype to distinguish bipolar from unipolar depression
evaluate the role played by confounding factors as psychotropic medications | 6 months
  evaluate the role played by confounding factors as psychotropic medications to distinguish bipolar from unipolar depression

CONTACTS AND LOCATIONS:
Overall Officials: jean Naudin, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Belzeaux R, Gorgievski V, Fiori LM, Lopez JP, Grenier J, Lin R, Nagy C, Ibrahim EC, Gascon E, Courtet P, Richard-Devantoy S, Berlim M, Chachamovich E, Theroux JF, Dumas S, Giros B, Rotzinger S, Soares CN, Foster JA, Mechawar N, Tall GG, Tzavara ET, Kennedy SH, Turecki G. GPR56/ADGRG1 is associated with response to antidepressant treatment. Nat Commun. 2020 Apr 2;11(1):1635. doi: 10.1038/s41467-020-15423-5. PMID 32242018